CLINICAL TRIAL: NCT01874379
Title: Investigating the Effect of the 'M'-Technique, Guided Imagery, or Standard of Care on Anxiety and Pain Pre- & Post-operatively in Elective Joint Replacement Patients.
Brief Title: 'M'-Technique, Guided Imagery, or Standard of Care on Anxiety and Pain Pre- & Post-operatively in Elective Joint Replacement Patients
Acronym: M•TIJRP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saint Clare's Health System (Other)
Collaborators: Saint Clare's Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M•TIJRP; WIRB #: 20121832 (Other: Western Institutional Review Board)
Record Dates: First submitted 2013-04-22; First posted 2013-06-11 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Hip or Knee Replacement
Keywords: Joint Replacement; Hip Replacement; Knee Replacement; Complementary Medicine Intervention
MeSH Terms: interventions — Imagery, Psychotherapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Guided Imagery (Experimental): The therapist will instruct the patient on the Guided Imagery protocol and will provide the patient with headphones and an MP-3 player to use for the guided imagery intervention. The patient will listen to the Guided Imagery for 18min 30 sec.
  Interventions: Other: Guided Imagery
- Standard of Care (Active Comparator): This group will serve as the control arm
  Interventions: Other: Standard of Care
- 'M'-Technique® (Experimental): The 'M'-Technique will be administered to the patient's hands and feet for a total of 18-20 minutes, to be equally divided between extremities used according to limitations as outlined. Any hand or foot that is accessed by an IV will be avoided.
  Interventions: Other: 'M'-Technique®

INTERVENTIONS:
Other: 'M'-Technique® — 'M'-Technique is a series of gentle stroking movements performed in a set sequence, with a set pressure of 3 on a scale of 0-10.
  Other Names: Light Structured Touch
  Arms: 'M'-Technique®
Other: Guided Imagery — Diane L. Tusek's Guided Imagery for Pre-Procedure/Surgery™ will be used.
  Arms: Guided Imagery
Other: Standard of Care — Normal Procedures, no complementary medicine intervention.
  Other Names: Control; No Intervention
  Arms: Standard of Care

SUMMARY:
In the M-TIJRP protocol the investigators will utilize two Integrative Medicine modalities in a randomized, controlled study using either the 'M'-Technique® developed by Jane Buckle, PhD or Diane L. Tusek's Guided Imagery for Pre-Procedure/Surgery™ with nature sounds to determine their effects on a specific group of pre- and post-operative patients, compared to no integrative medicine intervention - considered Standard of Care. A total of 225 patients undergoing surgical hip or knee replacement will participate; one third of the patient population will receive the 'M'-Technique touch intervention, one third will receive Tusek's Guided Imagery intervention delivered by headsets monitored by therapists from our Center for Complementary Medicine (CCM) and one third will comprise the control group, consisting of routine preoperative & postoperative care without integrated intervention.

Patients will be asked to complete Pain and Anxiety scales at four different timepoints throughout their hospital stay. These will occur at Same Day Surgery (pre-operatively), and Post Operatively Day 0, Day 1 & Day 2.

Rationale: Patients are often at their most vulnerable just prior to surgery when their stress and anticipation are high and again immediately afterward when their energy is lower and their bodies are trying to accommodate after an invasive procedure. In addition, the patient and his or her family sense a lack of control and feel a rise in anxiety over the possible outcomes. This stress, anxiety, and pain associated with surgery and recovery can increase complication rates and slow recovery times resulting in longer hospital stays.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Be receiving an initial or subsequent elective hip or knee replacement surgery

Exclusion Criteria:

1. Patients with an active infection or open wound in the location of the extremities where the 'M'-Technique will be performed
2. Patients with touch aversion
3. Non-English speaking patients - due to guided imagery recording availability in English only
4. Patients who demonstrate insufficient auditory discrimination as determined by their ability to engage in normal conversation
5. Patients who lack the sensation of being touched on the hands and/or feet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Symptomatic pain relief expressed in Visual Analogue Scales from no pain 0-10 worst possible pain | 18 months
  Measurement with Visual Analogue Scale
Symptomatic anxiety relief expressed in Visual Analogue Scales from no anxiety 0-10 worst possible anxiety | 18 months
  Visual Analogue Scale
Change from Baseline in Hamilton Anxiety Scale at Post Op Day 2 | 18 Months

SECONDARY OUTCOMES:
Patient Satisfaction Measure | 18 months
  Protocol specific questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: J. Brent Forward, MD, FACP, Principal Investigator — Saint Clare's Health System
Locations (1):
- Saint Clare's Health System, Denville, New Jersey, United States